CLINICAL TRIAL: NCT03543280
Title: Evaluation of the Value of Cerebral Perfusion Scintigraphy in the Study of Post-stroke Fatigability
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Other Study IDs: 6787
Record Dates: First submitted 2018-02-26; First posted 2018-06-01 (Actual); Last update posted 2018-06-01 (Actual); Status verified 2018-02

CONDITIONS: Fatigability Post Stroke
Keywords: fatigability post stroke; post stroke; high-speed CT; MRI

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
At present there is no consensus for post-stroke imaging except for the realization of early cerebral CT at 24 hours post-thrombolysis. The use of cerebral perfusion scintigraphy would predict the course of a stroke. Indeed, it has been shown that a good perfusion is linked to a good evolution of the neurological deficit. This test is used routinely to evaluate cerebral perfusion in patients with stroke. This technique was also used to study the mechanisms of post-stroke aphasia and to highlight neuronal disconnections after stroke, a reflection of the functioning of neural networks.

Neuropsychological tests are almost always done at 3 months. Fatigue is studied: PSF scale at 3 months, 6 months and 2 years. Research needs to be continued in this area because the pathophysiology remains unknown and the symptoms are disabling for patients. Using cerebral perfusion imaging would bring elements of understanding of this mechanism and ultimately improve the management of patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients: 18 to 60 years old at the initial diagnosis
* Admission for transient ischemic attack, stroke, dissection, TVC
* RANKIN less than or equal to 2
* Neuropsychological tests at +3 months: MoCA> 26 (to eliminate cognitive deteriorations too important for the good realization of the battery)
* Absence of psychiatric history
* Absence of psychotropic medication
* No history of stroke
* No complaint of pre-stroke fatigue
* Having signed the consent form

Exclusion Criteria:

* Impossibility of giving the subject or his family enlightened information (subject in emergency situation, difficulties in understanding the subject, etc.)
* Subject under the protection of justice
* Subject under guardianship or curatorship
* Refusal of the patient to participate in the study

Ages: 18 Years to 60 Years | Sex: All
Age Groups: Adult
Study Population: Patients with transient ischemic attack, stroke, dissection, TVC
Sampling Method: Probability Sample
Enrollment: 32 (Estimated)
Dates: Start 2018-02-23 (Actual); Primary Completion 2019-02 (Estimated); Study Completion 2019-02 (Estimated)

PRIMARY OUTCOMES:
Evaluate fatigue symptoms in stroke patients | After the period following a stroke: 1 month

CONTACTS AND LOCATIONS:
Locations (1):
- Service de Biophysique et de Médecine Nucléaire, Strasbourg, France

IPD SHARING:
Plan to Share IPD: No